CLINICAL TRIAL: NCT00632931
Title: A Randomized, Partially-Blind, Placebo-Controlled, 2-Period Crossover Study to Assess the Effects of a Single Dose of Vorinostat on the QTc Interval in Patients With Advanced Cancer
Brief Title: A Crossover Study to Assess the Effects of Vorinostat (MK0683, SAHA) in Patients With Advanced Cancer (0683-070)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0683-070; MK0683-070; 2008_515
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Cancer Relapsed; Advanced Cancer Refractory
MeSH Terms: interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- A (Experimental): Arm A: Drug/Placebo
  Interventions: Drug: vorinostat; Drug: Comparator: placebo (unspecified)
- B (Experimental): Arm B: Placebo/Drug
  Interventions: Drug: vorinostat; Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: vorinostat — A 2-part, crossover study. Part 1: Arm A: Single dose of vorinostat 800 mg capsules (Period 1) crossing over to Single dose of vorinostat Placebo capsules (Period 2) Arm B: Single dose of vorinostat Placebo capsules (Period 1) crossing over to Single dose of vorinostat 800 mg capsules (Period 2). Part 2: All patients will receive 400 mg vorinostat capsules once daily. Treatment will continue until disease progression or intolerable toxicity.
  Other Names: MK0683; Zolinza®
Drug: Comparator: placebo (unspecified) — A 2-part, crossover study. Part 1: Arm A: Single dose of vorinostat Placebo capsules (Period 2) Arm B: Single dose of vorinostat Placebo capsules (Period 1).

SUMMARY:
A 2-period, crossover study to assess the effects of MK0683 (vorinostat) on the QTc interval in patients with relapsed or refractory advanced cancer.

DETAILED DESCRIPTION:
Merck Duration of Treatment : vorinostat; treatment will continue until disease progression or intolerable toxicity is reached

ELIGIBILITY:
Inclusion Criteria:

* Patient has a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy or for which standard therapy does not exist
* Patient has life expectancy of greater than 3 months
* Patient is able to swallow capsules

Exclusion Criteria:

* Patient has had chemotherapy, radiotherapy or biological therapy 2 weeks prior to taking study drug
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent
* Patient has active CNS metastases and/or carcinomatous meningitis
* Patient has primary central nervous system tumor
* Patient has a history of drug or alcohol abuse
* Patient has Hepatitis B or C
* Patient is HIV positive
* Patient has active infection or has received intravenous antibiotics, antiviral or antifungal agents 2 weeks before taking study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Munster PN, Rubin EH, Van Belle S, Friedman E, Patterson JK, Van Dyck K, Li X, Comisar W, Chodakewitz JA, Wagner JA, Iwamoto M. A single supratherapeutic dose of vorinostat does not prolong the QTc interval in patients with advanced cancer. Clin Cancer Res. 2009 Nov 15;15(22):7077-84. doi: 10.1158/1078-0432.CCR-09-1214. Epub 2009 Nov 3. PMID 19887475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eric Rubin, M.D., The Cancer Institute of New Jersey, New Brunswick, New Jersey; Pamela Munster, M.D., H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida; Prof. Dr. Simon van Belle, University Hospital of Ghent, Ghent, Belgium.
  Dosing initiated on 16-Jul-2007 and completed on 05-Feb-2009.
Pre-assignment Details: Enrolled patients were assigned to 1 of 2 dose sequences (vorinostat then placebo or placebo then vorinostat) in Part 1 of the study to determine the effect of vorinostat on the QTcF (Fridericia-corrected QT) interval. Following Part 1, active patients continued into Part 2, daily dosing of vorinostat.
Groups:
- Vorinostat Then Placebo: Part 1: Single dose 800 mg vorinostat in Period 1 followed by a three day wash out period, then matching placebo in Period 2. Following the last dose of study drug, there was a minimum 5 day washout before entering Part 2.
- Placebo Then Vorinostat: Part 1: Single dose matching placebo in Period 1 followed by a three day wash out period, then single dose 800 mg vorinostat in Period 2. Following the last dose of study drug, there was a minimum 5 day washout before entering Part 2.
- All Participants: Part 2: Vorinostat 400 mg once daily.
  Ten participants changed dosage to vorinostat 300 mg daily during Part 2.
Period: Part 1, Period 1
Arm/Group | Vorinostat Then Placebo: Part 1 | Placebo Then Vorinostat: Part 1 | All Participants: Part 2
Started | 13 | 12 | 0
Completed | 11 | 12 | 0
Not Completed | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part 1, Washout
Arm/Group | Vorinostat Then Placebo: Part 1 | Placebo Then Vorinostat: Part 1 | All Participants: Part 2
Started | 11 | 12 | 0
Completed | 11 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Part 1, Period 2
Arm/Group | Vorinostat Then Placebo: Part 1 | Placebo Then Vorinostat: Part 1 | All Participants: Part 2
Started | 11 | 12 | 0
Completed | 11 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Post-Part 1 Washout
Arm/Group | Vorinostat Then Placebo: Part 1 | Placebo Then Vorinostat: Part 1 | All Participants: Part 2
Started | 12 (1 patient who did not complete Period 1 was subsequently enrolled into Post Part 1) | 12 | 0
Completed | 12 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Part 2
Arm/Group | Vorinostat Then Placebo: Part 1 | Placebo Then Vorinostat: Part 1 | All Participants: Part 2
Started | 0 | 0 | 24
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 24
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Participants group includes data from all participants throughout Part 1 and Part 2 of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 59.4 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black | 2
  Hispanic | 1
  White | 21
Cancer Type [Number; unit: Participants]
  Ovarian | 5
  Colon | 3
  Lung | 3
  Mesothelioma | 3
  Uterine | 2
  Soft Tissue | 2
  Anal | 1
  Basocellular | 1
  Breast | 1
  Gastrointestinal | 1
  Mucinous carcinoma | 1
  Pancreatic | 1
  Thyroid | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG Scale: 0 = Normal Activity, 1 = Symptoms, but ambulatory, 2 = In bed <50% of the time, 3 = In bed >50% of the time, 4 = 100% Bedridden, 5 = Dead
  Participants
    0 = Normal Activity | 9
    1 = Symptoms, but ambulatory | 13
    2 = In bed <50% of the time | 3
Number of Prior Radiation Therapies [Number; unit: Participants]
  None | 14
  One Prior Radiation Therapy | 7
  Two Prior Radiation Therapies | 1
  Three or More Prior Radiation Therapies | 3
Number of Prior Systemic Anti-Cancer Therapies [Number; unit: Participants]
  One Prior Systemic Anti-Cancer Therapy | 0
  Two Prior Systemic Anti-Cancer Therapies | 3
  Three or more Prior Systemic Anti-Cancer Therapies | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QTcF at 0.5 Hours
Description: The Fridericia correction of the QT interval (QTcF) was determined at each time point from five replicate measurements. The change from baseline in QTcF was calculated by subtracting the QTcF value at each timepoint from the QTcF baseline (predose) value.
Time Frame: Baseline and 0.5 hours
Population: All patients as treated population in Part 1 of the Study;
  22 patients had QTcF data from the vorinostat period (One patient with protocol violation, and two patients without predose measurements were excluded) and 23 patients had QTcF data from the placebo period (one patient with protocol violation and one patient who discontinued were excluded)
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 22
milliseconds | 1.78 [-1.53 to 5.09] | -1.22 [-4.53 to 2.08]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 3.00, 90% CI [-0.28 to 6.28]

2. Primary Outcome: Change From Baseline in QTcF at 1 Hour
Description: Fridericia correction of the QT interval (QTcF) was determined at each time point from five replicate measurements. The change from baseline in QTcF was calculated by subtracting the QTcF value at each timepoint from the QTcF baseline (predose) value.
Time Frame: Baseline and 1 hour
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 22
milliseconds | 0.22 [-3.09 to 3.52] | -1.23 [-4.54 to 2.08]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 1.45, 90% CI [-1.38 to 4.72]

3. Primary Outcome: Change From Baseline in QTcF at 2 Hours
Description: as for outcome 1
Time Frame: Baseline and 2 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds | 1.09 [-2.22 to 4.40] | -1.98 [-5.23 to 1.28]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 3.07, 90% CI [-0.17 to 6.31]

4. Primary Outcome: Change From Baseline in QTcF at 3 Hours
Description: as for outcome 1
Time Frame: Baseline and 3 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds | 1.32 [-1.99 to 4.63] | -1.52 [-4.77 to 1.73]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 2.84, 90% CI [-0.40 to 6.08]

5. Primary Outcome: Change From Baseline in QTcF at 4 Hours
Description: The Fridericia correction of the QT interval (QTcF) was determined at each time point from five replicate measurements. The placebo-corrected change from baseline in QTcF was calculated by subtracting the QTcF change from baseline for placebo at each timepoint from the QTcF change from baseline for vorinostat at each timepoint.
Time Frame: Baseline and 4 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds | 4.95 [1.64 to 8.26] | -1.49 [-4.75 to 1.76]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 6.44, 90% CI [3.21 to 9.68]

6. Primary Outcome: Change From Baseline in QTcF at 8 Hours
Description: as for outcome 1
Time Frame: Baseline and 8 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 23 | 22
milliseconds | -3.56 [-6.87 to -0.25] | -7.89 [-11.20 to -4.58]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 4.33, 90% CI [1.05 to 7.60]

7. Primary Outcome: Change From Baseline in QTcF at 12 Hours
Description: as for outcome 1
Time Frame: Baseline and 12 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 21 | 22
milliseconds | 1.35 [-2.08 to 4.78] | -1.31 [-4.62 to 2.00]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 2.66, 90% CI [-0.70 to 6.02]

8. Primary Outcome: Change From Baseline in QTcF at 24 Hours
Description: as for outcome 1
Time Frame: Baseline and 24 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Vorinostat | Placebo
Number analyzed (Participants) | 22 | 22
milliseconds | 1.53 [-1.84 to 4.98] | -4.89 [-8.29 to -1.67]
Statistical Analysis 1: Comparison: Vorinostat vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 6.51, 90% CI [3.19 to 9.82]

ADVERSE EVENTS:
Time Frame: Reported adverse experiences are those from the time patients began study treatment until the patient discontinued. The average AE reporting timeframe is 78 days.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=25)
Anemia (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Disease Progression (General disorders) | 3
Fatigue (General disorders) | 1
Pyrexia (Gastrointestinal disorders) | 2
Portal Vein Thrombosis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=25)
Anemia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Dry Eye (Eye disorders) | 1
Abdominal Cramp (Gastrointestinal disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Fullness (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 9
Dry Mouth (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gas (Gastrointestinal disorders) | 1
Gas Pain (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Loose Stools (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 10
Axillary Pain (General disorders) | 1
Chest Pain (General disorders) | 2
Chills (General disorders) | 1
Early Satiety (General disorders) | 2
Fatigue (General disorders) | 17
Fever (General disorders) | 2
Foot Edema (General disorders) | 1
Gait Unsteady (General disorders) | 1
Intermittent Pyrexia (General disorders) | 1
Leg Edema (General disorders) | 1
Edema Lower Limb (General disorders) | 1
Suprapubic Pain (General disorders) | 1
Weakness (General disorders) | 1
Weakness Generalized (General disorders) | 1
Candidiasis (Infections and infestations) | 1
Sinus Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 3
Wound Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alkaline Phosphatase Increased (Investigations) | 3
Blood Bilirubin Increased (Investigations) | 1
Blood Carbon Dioxide Increased (Investigations) | 1
Blood Creatine Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 2
Blood Glucose Increased (Investigations) | 1
Blood Magnesium Decreased (Investigations) | 1
Blood Magnesium Increased (Investigations) | 2
Blood Potassium Decreased (Investigations) | 2
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 1
International Normalized Ratio Increased (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
Prothrombin Time Prolonged (Investigations) | 1
Skin Turgor Decreased (Investigations) | 1
Weight Decreased (Investigations) | 4
White Blood Cell Count Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Decreased Appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hyperchloremia (Metabolism and nutrition disorders) | 1
Hypercreatininemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperphosphatasemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Foot Cramps (Musculoskeletal and connective tissue disorders) | 1
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Hip (Musculoskeletal and connective tissue disorders) | 2
Pain In Leg (Musculoskeletal and connective tissue disorders) | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3
Unilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 1
Neuropathic Pain (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Numbness (Nervous system disorders) | 1
Numbness In Toes (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Taste Changed (Nervous system disorders) | 6
Tingling (Nervous system disorders) | 1
Tingling Feet/Hands (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Bladder Discomfort (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Urine Discoloration (Renal and urinary disorders) | 1
Benign Prostatic Hypertrophy (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Spotting Vaginal (Reproductive system and breast disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Inferior Venacaval Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.